CLINICAL TRIAL: NCT02265484
Title: A Randomized Open Labelled Placebo Controlled Trial to Study the Efficacy of Bromocriptine in Patients With Hepatic/Cirrhosis Related Parkinsonism
Brief Title: To Study the Efficacy of Bromocriptine in Patients With Hepatic/Cirrhosis Related Parkinsonism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-bromocriptine-01
Record Dates: First submitted 2014-09-12; First posted 2014-10-16 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2013-04

CONDITIONS: Cirrhosis Related Parkinsonism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactulose + Rifaximin + Bromocriptine (Experimental)
  Interventions: Drug: Lactulose+Rifaximin +Bromocriptine
- Lactulose+Rifaximin+Placebo (Active Comparator)
  Interventions: Drug: Lactulose+Rifaximin +Bromocriptine

INTERVENTIONS:
Drug: Lactulose+Rifaximin +Bromocriptine

SUMMARY:
After successful screening of liver cirrhosis patients attending ILBS OPD for signs of parkinsonism ( tremor, rigidity or bradykinesia, any 2 of 3). Diagnosis of hepatic/cirrhosis related parkinsonism will be made. Patients will be randomized into Bromocriptine and Placebo. Patients will be followed up every month in OPD (Out Patient Department), ILBS (Institute of liver & Biliary Sciences) for 3 months. Detailed neurological examination will be done at each visit & UPDRS (Unified Parkinson's Disease Rating Scale ) score will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis of liver with signs of parkinsonisms
* Patients consented for the study protocol by signing the informed consent.

Exclusion Criteria:

* Age < 18 years.
* Patient s with HCC (Hepatocellular Carcinoma).
* Patients diagnosed as Wilsons disease.
* Patient who withdrew or non complaint to the study protocol.
* ALF (Acute Liver failure)
* Classical Parkinsonism
* Atypical Parkinsonism
* Pregnancy
* Hypotension
* Uncontrolled hypertension
* CAD
* Psychiatric illness
* Acute episode of Hepatic encephlopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be decrement in UPDRS (Unified Parkinson's Disease Rating Scale) score by 30 %. | 3 months

SECONDARY OUTCOMES:
The secondary end point will be decrement in UPDRS (Unified Parkinson's Disease Rating Scale) score of 10% to 30%. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Amrish Sahney, MD, Principal Investigator — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Sahney A, Sharma BC, Jindal A, Anand L, Arora V, Vijayaraghavan R, Dhamija RM, Kumar G, Bhardwaj A, Sarin SK. A double-blind randomized controlled trial to assess efficacy of bromocriptine in cirrhotic patients with hepatic parkinsonism. Liver Int. 2019 Apr;39(4):684-693. doi: 10.1111/liv.14024. Epub 2019 Feb 4. PMID 30554466